CLINICAL TRIAL: NCT02180971
Title: Diagnostic Usefulness of Multidetector Coronary CT in Vasospastic Angina
Brief Title: Multidetector Coronary CT In Vasospastic Angina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, M.D. Director, Regional Clinical Trial Center. Professor, Dept. of Cardiology Dong-A Unicersity Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DOMINATION
Record Dates: First submitted 2014-06-29; First posted 2014-07-03 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Vasospastic Angina
Keywords: Multi-detector computed tomography angiography; Coronary vessel distensibility; Coronary spasm
MeSH Terms: conditions — Angina Pectoris, Variant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive CAG with EG test (Experimental): A positive finding for coronary angiography with an ergonovine provocation test is defined as transient, total, or sub-total occlusion (>90% stenosis) with signs/symptoms of myocardial ischemia (chest pain and ischemic ECG change).
  Interventions: Procedure: Positive CAG with EG test
- Negative CAG with EG test (Experimental): Negative test: less than 70% luminal narrowing, without chest pain or ST-segment changes after ergonovine coronary injection
  Interventions: Procedure: Negative CAG with EG test

INTERVENTIONS:
Procedure: Positive CAG with EG test — A positive finding for coronary angiography with an ergonovine provocation test is defined as transient, total, or sub-total occlusion (>90% stenosis) with signs/symptoms of myocardial ischemia (chest pain and ischemic ECG change).
  Arms: Positive CAG with EG test
Procedure: Negative CAG with EG test — Negative test: less than 70% luminal narrowing, without chest pain or ST-segment changes after ergonovine coronary injection
  Arms: Negative CAG with EG test

SUMMARY:
The purpose of this study is to compare the extent of coronary vessel stenosis between coronary spasm-induced angina attacks (named vasospastic angina, VSA) patients and health volunteers by multi-detector computed tomography angiography (MDCTA), and to evaluate the diagnostic efficacy of MDCTA in patients with VSA.

DETAILED DESCRIPTION:
Vasospastic angina (VSA) was characterized by transient ischemic ST-segment change during angina attacks. Coronary spasm provocation test, as a diagnostic golden standard, has been widely used for the management of VSA according to JCS 2013 guidelines.

With regard to the characteristics of spasm segment, had been clearly described by other invasive imaging methods including intravascular ultrasound and optical coherence tomography. However, there is potential risk during these invasive procedures, such as severe myocardial ischemia or fatal arrhythmia.

Presently available imaging test for coronary artery disease including multi-detector computed tomography angiography (MDCTA) with high diagnostic accuracy to evaluate coronary artery stenosis. However, the diagnostic accuracy of MDCTA in patients with VSA is lacking.

Therefore, more efficient and safe noninvasive diagnostic method is required for the detection of angina-like attacks patients.

ELIGIBILITY:
Inclusion Criteria:

* Onset of angina-like attack at rest, during effort, or during rest and effort.
* Patients will be scheduled to undergo multi-detector computed tomography angiography and coronary angiography with an ergonovine provocation test.

Exclusion Criteria:

* Evidence of acute coronary syndrome, cardiomyopathy and valvular heart disease.
* More than 50% stenosis detected by coronary angiography .
* Renal insufficiency (serum creatine>2.5 mg/dl).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Characteristics of coronary lesion | CAG will be performed after multidetector coronary CT, an expected average of 4 weeks.
  1. Plaque composition: noncalcified plaque, which is < 130 Hounsfield units(HU). Calcified plaque with a density of > 130 HU. Mixed plaque: plaque area consisted of > 50% of non-calcified plaque.
  2. The remodeling index (RI) was calculated by dividing the cross-sectional lesion vessel-area by the reference vessel area.Positive remodeling was defined as RI > 1.05, otherwise RI ≤0.95.
  3. Significant stenosis is defined as stenosis in more than 50% of the coronary artery diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, M.D., Principal Investigator — Dong-A University Hospital, Busan, Republic of Korea
Locations (1):
- DongA University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kang KM, Choi SI, Chun EJ, Kim JA, Youn TJ, Choi DJ. Coronary vasospastic angina: assessment by multidetector CT coronary angiography. Korean J Radiol. 2012 Jan-Feb;13(1):27-33. doi: 10.3348/kjr.2012.13.1.27. Epub 2011 Dec 23. PMID 22247633
- [Result] Ghersin E, Litmanovich D, Dragu R, Rispler S, Lessick J, Ofer A, Brook OR, Gruberg L, Beyar R, Engel A. 16-MDCT coronary angiography versus invasive coronary angiography in acute chest pain syndrome: a blinded prospective study. AJR Am J Roentgenol. 2006 Jan;186(1):177-84. doi: 10.2214/AJR.04.1232. PMID 16357399
- [Result] JCS Joint Working Group. Guidelines for diagnosis and treatment of patients with vasospastic angina (Coronary Spastic Angina) (JCS 2013). Circ J. 2014;78(11):2779-801. doi: 10.1253/circj.cj-66-0098. Epub 2014 Sep 30. No abstract available. PMID 25273915
- [Result] Tsujita K, Sakamoto K, Kojima S, Kojima S, Takaoka N, Nagayoshi Y, Sakamoto T, Tayama S, Kaikita K, Hokimoto S, Sumida H, Sugiyama S, Nakamura S, Ogawa H. Coronary plaque component in patients with vasospastic angina: a virtual histology intravascular ultrasound study. Int J Cardiol. 2013 Oct 3;168(3):2411-5. doi: 10.1016/j.ijcard.2013.02.002. Epub 2013 Feb 27. PMID 23453453
- [Result] Morikawa Y, Uemura S, Ishigami K, Soeda T, Okayama S, Takemoto Y, Onoue K, Somekawa S, Nishida T, Takeda Y, Kawata H, Horii M, Saito Y. Morphological features of coronary arteries in patients with coronary spastic angina: assessment with intracoronary optical coherence tomography. Int J Cardiol. 2011 Feb 3;146(3):334-40. doi: 10.1016/j.ijcard.2009.07.011. Epub 2009 Aug 27. PMID 19716193